CLINICAL TRIAL: NCT04639908
Title: Federal Knowledge Centre for Health Care
Acronym: KCEHR2020-02
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: KCE
Record Dates: First submitted 2020-10-23; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Integrated Care
Keywords: elderly care; primary care; belgium
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- barriers: find out what are the barriers
  Interventions: Other: Interview
- facilitators: find out what are the facilitators
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — interview with patient

SUMMARY:
In order to prepare for the ageing population and its impact on the health care system, the National Institute for Sickness and Disability Insurance in Belgium (RIZIV) launched in 2010 a subsidy programme (called Protocol 3) for innovative projects aimed at care and support for vulnerable older people with complex care needs. The objective of these projects is to reduce the risk and need for admission to a care institution/residential care centre. These are alternative and supportive forms of care for the elderly for which there is currently no allowance, which enable vulnerable older people to be cared for at home, which have a positive influence on the evolution of the older person's state of health and which improve the quality of life, which do not entail higher costs than those of a classic admission and which are scientifically evaluated.

These Protocol 3 projects focus on vulnerable elderly people who are not admitted to a residential care centre, but who are at risk of a complex and/or long-term care situation. As a result of the complex care situation, there is also a great need for coordinated care between different care providers and/or there will also be supportive forms of care that ensure continuity of care. The expected added value of the care innovation projects should focus on: the importance of consultation and cooperation between the various stakeholders, the means to improve the competences of all relevant stakeholders, the means to organise customised care and the means to achieve continuity of care for the patient. The objective of the current study is to evaluate the phase 2 interventions, in particular: the adapted interventions case management and occupational therapy; and the newly introduced interventions in phase 3: health education, educational sessions for informal care providers and control visits at night.

DETAILED DESCRIPTION:
In order to prepare for the ageing population and its impact on the health care system, the National Institute for Sickness and Disability Insurance in Belgium (RIZIV) launched in 2010 a subsidy programme (called Protocol 3) for innovative projects aimed at care and support for vulnerable older people with complex care needs. The objective of these projects is to reduce the risk and need for admission to a care institution/residential care centre. These are alternative and supportive forms of care for the elderly for which there is currently no allowance, which enable vulnerable older people to be cared for at home, which have a positive influence on the evolution of the older person's state of health and which improve the quality of life, which do not entail higher costs than those of a classic admission and which are scientifically evaluated.

These Protocol 3 projects focus on vulnerable elderly people who are not admitted to a residential care centre, but who are at risk of a complex and/or long-term care situation. As a result of the complex care situation, there is also a great need for coordinated care between different care providers and/or there will also be supportive forms of care that ensure continuity of care. The expected added value of the care innovation projects should focus on: the importance of consultation and cooperation between the various stakeholders, the means to improve the competences of all relevant stakeholders, the means to organise customised care and the means to achieve continuity of care for the patient. The objective of the current study is to evaluate the phase 2 interventions, in particular: the adapted interventions case management and occupational therapy; and the newly introduced interventions in phase 3: health education, educational sessions for informal care providers and control visits at night.

After all, an evaluation at the end of these projects is important in order to evaluate the added value of these care innovation projects and how they can possibly be structurally anchored. The starting point of this study is to learn in a qualitative way about the perceptions and experiences of patients and their informal carers about the benefits of the interventions, the barriers and facilitating factors of their implementation and the potential for improvement of these initiatives. The objective is to assess the extent to which patient needs are met by the interventions and what can be improved to consolidate the intervention or add more value to it.

ELIGIBILITY:
Inclusion Criteria:

* uses interventions of protocol 3 projects

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who profit from the interventions offered by Protocol 3
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-04-09 (Estimated); Study Completion 2021-04-09 (Estimated)

PRIMARY OUTCOMES:
incidence of falling at home | 8 months
  interview
admission in nursing home | 8 months
  interview

CONTACTS AND LOCATIONS:
Overall Officials: Justien Cornelis, PhD, Principal Investigator — KCE

IPD SHARING:
Plan to Share IPD: No